CLINICAL TRIAL: NCT03354598
Title: A Prospective Phase 3 Randomized Multi-center Double-blind Study of Efficacy Tolerability & Safety of Oral Sulopenem-etzadroxil/Probenecid vs Ciprofloxacin for Treatment of Uncomplicated Urinary Tract Infections (uUTI) in Adult Women
Brief Title: Oral Sulopenem-etzadroxil/Probenecid Versus Ciprofloxacin for Uncomplicated Urinary Tract Infection in Adult Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT001-301
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2019-12

CONDITIONS: Uncomplicated Urinary Tract Infections
MeSH Terms: interventions — Probenecid; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulopenem-etzadroxil/probenecid (Experimental): Sulopenem-etzadroxil/probenecid 500 mg PO twice daily for 5 days
  Interventions: Drug: Sulopenem-Etzadroxil/Probenecid
- Ciprofloxacin (Active Comparator): Ciprofloxacin 250 mg PO administered twice daily for 3 days
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Sulopenem-Etzadroxil/Probenecid — Treatment of uncomplicated urinary tract infection
  Arms: Sulopenem-etzadroxil/probenecid
Drug: Ciprofloxacin — Treatment of uncomplicated urinary tract infection
  Other Names: Cipro
  Arms: Ciprofloxacin

SUMMARY:
This is a prospective, Phase 3, randomized, multi-center, double-blind study of the efficacy, tolerability, and safety of oral sulopenem-etzadroxil/probenecid versus oral ciprofloxacin for treatment of uncomplicated urinary tract infection (uUTI) in adult women

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥18 years of age with 24-96 hours of urinary symptoms attributable to a urinary tract infection (UTI)
2. Two of the following signs and symptoms of uUTI: urinary frequency, urinary urgency, pain or burning micturition, suprapubic pain
3. A mid-stream urine specimen with:

   1. a dipstick analysis positive for nitrite AND
   2. evidence of pyuria as defined by either:

   i. a dipstick analysis positive for leukocyte esterase ii. at least 10 white blood cells per cubic millimeter on microscopic analysis of unspun urine iii. White blood cell count ≥10 cells/high-powered field in the sediment of a spun urine
4. Has given written informed consent to participate in the study.

Exclusion Criteria:

1. Presence of signs and symptoms suggestive of acute pyelonephritis: fever (temperature > 38°Celsius), chills, costovertebral angle tenderness, flank pain, nausea, and/or vomiting
2. Receipt of antibacterial drug therapy potentially effective as treatment of uUTI within the prior 7 days
3. Concurrent use of non-study treatments that would have a potential effect on outcome evaluations in patients with uUTI
4. Patients with ileal loops or urinary stoma
5. Patients with an indwelling urinary catheter in the previous 30 days
6. Patients with paraplegia
7. Patients who are likely to receive ongoing antibacterial drug prophylaxis after treatment of uUTI (e.g., patients with vesico-ureteral reflux)
8. Any history of trauma to the pelvis or urinary tract
9. Patient's urine culture, if available at study entry, identify more than 2 microorganisms regardless of colony count or patient has a confirmed fungal UTI
10. Patient is receiving hemodialysis or peritoneal dialysis or had a renal transplant
11. Known history of creatinine clearance <50 mL/min
12. Patients known to have liver disease
13. Patients who are pregnant, or females of child-bearing age unable to take adequate contraceptive precautions
14. Patients with uncontrolled diabetes mellitus
15. Patients with history of blood dyscrasias
16. Patients with history of uric acid kidney stones
17. Patients with acute gouty attack
18. Patients on chronic methotrexate therapy
19. Patient known to be immunocompromised
20. Patients with a known history of myasthenia gravis
21. Patients who require concomitant administration of tizanidine or valproic acid
22. Patients with a history of allergy or hypersensitivity to carbapenems, beta-lactams, quinolones or probenecid
23. Patient is considered unlikely to survive the 4-week study period or has a rapidly progressive or terminal illness including septic shock which is associated with a high risk of mortality
24. History of seizures
25. Use of any other investigational drug in the 30 days prior to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are eligible for this study.
Enrollment: 1671 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Medical Facility, Birmingham, Alabama
  - Medical Facility, Phoenix, Arizona
  - Medical Facility, Tolleson, Arizona
  - Medical Facility, Cerritos, California
  - Medical Facility, Chula Vista, California
  - Medical Facility, Fullerton, California
  - Medical Facility, La Mesa, California
  - Medical Facility, Los Angeles, California
  - Medical Facility, San Diego, California
  - Medical Facility, Sylmar, California
  - Medical Facility, Washington D.C., District of Columbia
  - Medical Facility, Bradenton, Florida
  - Medical Facility, Clearwater, Florida
  - Medical Facility, Doral, Florida
  - Medical Facility, Edgewater, Florida
  - Medical Facility, Hialeah, Florida
  - Medical Facility, Lauderdale Lakes, Florida
  - Medical Facility, Miami, Florida
  - Medical Facility, Miami Springs, Florida
  - Medical Facility, New Port Richey, Florida
  - Medical Facility, Ormond Beach, Florida
  - Medical Facility, Palmetto Bay, Florida
  - Medical Facility, St. Petersburg, Florida
  - Medical Facility, Winter Haven, Florida
  - Medical Facility, Atlanta, Georgia
  - Medical Facility, Norcross, Georgia
  - Medical Facility, Perry, Georgia
  - Medical Facility, Lake Charles, Louisiana
  - Medical Facility, Metairie, Louisiana
  - Medical Facility, New Orleans, Louisiana
  - Medical Facility, Las Vegas, Nevada
  - Medical Facility, Brooklyn, New York
  - Medical Facility, Raleigh, North Carolina
  - Medical Facility, Hugo, Oklahoma
  - Medical Facility, Easley, South Carolina
  - Medical Facility, Lancaster, South Carolina
  - Medical Facility, Myrtle Beach, South Carolina
  - Medical Facility, Austin, Texas
  - Medical Facility, Carrollton, Texas
  - Medical Facility, Corpus Christi, Texas
  - Medical Facility, Dallas, Texas
  - Medical Facility, Houston, Texas
  - Medical Facility, Pearland, Texas
  - Medical Facility, Plano, Texas
  - Medical Facility, Sugar Land, Texas
  - Medical Facility, Bountiful, Utah
  - Medical Facility, Salt Lake City, Utah
  - Medical Facility, South Jordan, Utah
  - Medical Facility, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunne MW, Aronin SI, Das AF, Akinapelli K, Zelasky MT, Puttagunta S, Boucher HW. Sulopenem or Ciprofloxacin for the Treatment of Uncomplicated Urinary Tract Infections in Women: A Phase 3, Randomized Trial. Clin Infect Dis. 2023 Jan 6;76(1):66-77. doi: 10.1093/cid/ciac738. PMID 36069202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulopenem-etzadroxil/Probenecid | Ciprofloxacin
Started | 835 | 836
Microbiologic Modified Intent to Treat Resistant (Micro-MITTR) Participants | 147 | 139
Microbiologic Modified Intent to Treat Susceptible (Micro-MITTS) Participants | 370 | 415
Microbiologic Modified Intent to Treat (Micro-MITT) Participants | 517 | 554
Modified Intent to Treat (MITT) Participants | 785 | 794
Intent to Treat (ITT) Participants | 787 | 803
Safety Participants | 833 | 827
Completed | 755 | 761
Not Completed | 80 | 75

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulopenem-etzadroxil/Probenecid | Ciprofloxacin | Total
Number analyzed (Participants) | 787 | 803 | 1590
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (18.8) | 50.0 (19.1) | 49.9 (19.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 787 | 803 | 1590
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 253 | 232 | 485
  Not Hispanic or Latino | 529 | 570 | 1099
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 448 | 441 | 889
  Ukraine | 144 | 137 | 281
  Russia | 195 | 225 | 420
Diabetes [Count of Participants; unit: Participants] | 93 | 106 | 199

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Microbiologic Modified Intent to Treat Resistant (Micro-MITTR) Participants With Overall Success
Description: Overall Success: Clinical Success (resolution of uncomplicated urinary tract infection (uUTI) symptoms present at study entry and no new symptoms) AND Microbiologic success (eradication of the baseline pathogen)
Time Frame: Day 12+/-1 day
Population: micro-MITTR population: patients with baseline uropathogen non-susceptible to the comparator ciprofloxacin.
Measure: Number; unit: percentage of participants
Arm/Group | Sulopenem-etzadroxil/Probenecid | Ciprofloxacin
Number analyzed (Participants) | 147 | 139
percentage of participants | 62.6 | 36.0

2. Primary Outcome: Percentage of Microbiologic Modified Intent to Treat Susceptible (Micro-MITTS) Participants With Overall Success
Description: Overall Success is Clinical Success (resolution of uUTI symptoms present at study entry and no new uUTI symptoms) AND Microbiologic success (eradication of the baseline pathogen)
Time Frame: Day 12 +/- 1 day
Population: micro-MITTS population: patients with baseline uropathogen susceptible to the comparator ciprofloxacin.
Measure: Number; unit: percentage of participants
Arm/Group | Sulopenem-etzadroxil/Probenecid | Ciprofloxacin
Number analyzed (Participants) | 370 | 415
percentage of participants | 66.8 | 78.6

3. Secondary Outcome: Percentage of Microbiologic Modified Intent to Treat Resistant (Micro-MITTR) Patients With Microbiologic Success
Description: Microbiologic success is defined as eradication of the baseline pathogen (<1000 Colony Forming Units (CFU)/mL) at the Test of Cure visit
Time Frame: Day 12+/-1 day
Population: micro-MITTR population: patients with baseline uropathogen non-susceptible to the comparator ciprofloxacin.
Measure: Number; unit: percentage of participants
Arm/Group | Sulopenem-etzadroxil/Probenecid | Ciprofloxacin
Number analyzed (Participants) | 147 | 139
percentage of participants | 74.1 | 49.6

4. Other Pre Specified Outcome: Percentage of Microbiologic Modified Intent to Treat (Micro-MITT) Participants With Overall Success
Description: as for outcome 2
Time Frame: 12 +/- 1 day
Population: micro-MITT population: micro-MITTR and micro-MITTS (ciprofloxacin nonsusceptible and ciprofloxacin susceptible) populations combined.
Measure: Number; unit: percentage of participants
Arm/Group | Sulopenem-etzadroxil/Probenecid | Ciprofloxacin
Number analyzed (Participants) | 517 | 554
percentage of participants | 65.6 | 67.9

ADVERSE EVENTS:
Time Frame: From the time of informed consent through the final visit, an average of 28 days.
Arm/Group | Sulopenem-etzadroxil/Probenecid | Ciprofloxacin
All-Cause Mortality (participants affected / at risk) | 1/833 | 0/827
Serious Adverse Events (participants affected / at risk) | 6/833 | 2/827
Other Adverse Events (participants affected / at risk) | 103/833 | 21/827
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulopenem-etzadroxil/Probenecid (N=833) | Ciprofloxacin (N=827)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
small intestine obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
chest pain (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
urosepsis (Infections and infestations) | 1 (1) | 0 (0)
lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
presuncope (Nervous system disorders) | 1 (1) | 0 (0)
angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulopenem-etzadroxil/Probenecid (N=833) | Ciprofloxacin (N=827)
Diarrhea (Gastrointestinal disorders) | 103 (947) | 21 (91)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will provide Iterum opportunity to review proposed publication/other type of disclosure before submitted/disclosed. PI will provide full text of intended disclosure to Iterum at least 30 days before submitted/disclosed. If any patent action is required to protect intellectual property rights, PI agrees to delay disclosure for a period not to exceed an additional 60 days. PI will, on request, remove previously undisclosed Confidential Information before disclosure.

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT03354598/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT03354598/SAP_001.pdf